CLINICAL TRIAL: NCT05734131
Title: Phenotyping Knee Osteoarthritis Patients According to Patient's Pain Experience and Its Correlation Between Gait Parameters and Time Up&Go Test: an Observational Study
Brief Title: Biopsychosocial Assessment in Knee OA
Acronym: BioPsyOA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: FDG_biopsycho_OA
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bio-psychosocial assessment — Kinematic parameters were analyzed by two functional tests, the 10-Meter Walking Test (10MWT) and the Time Up&Go test (TUG).
  Other Names: 10MWT and TUG test

SUMMARY:
Background: Patient's pain experience is a complex phenomenon. A comprehensive clinical assessment of the patient's pain experience is helpful to define individual differences between patients and thus to plan effective individualized treatment programs. Gait assessment is an important functional task in the clinical evaluation, which allows the definition and modulation of therapeutic intervention. The influence of patient's pain experience on gait parameters is currently understudied in literature.

Objective: To investigate patient's pain experience based on an assessment model proposed by Walton and Elliott in patients with knee OA. The study's second aim is to examine the correlation between the parameters of the 10 Meter Walking Test (10MWT) and Time Up and Go test (TUG) assessed by an inertial sensor and the patient's pain experience.

DETAILED DESCRIPTION:
Each patient undergoes a clinical pain assessment including Western Ontario and McMaster University Osteoarthritis (WOMAC) scale, a patient-reported outcome questionnaire that aims to identify changes in symptoms and activity restrictions in subjects with OA. A guided clinical assessment explores nociceptive, neuropathic, nociplastic, psychological, beliefs, socioenvironmental, and sensorimotor disintegration domains. A series of assessment scales were considered for each patient: Pain DETECT Scale; Central Sensitization Inventory (CSI) Index; Patient Health Questionairre (PHQ-9); post traumatic distress checklist (PTSD); Pain Catastrophyzing Scale (PCS); Tampa Kinesiophobia Scale (TSK); Fear Avoidance Believe Questionnaire (FABQ), Injustice Experience Questionnaire (IEQ) and the completion of a body chart.

An assessment of pressure pain threshold (PPT) was conducted through an electronic algometer (Algomed). The defined sites for PPT were the patella, Gerdy's tubercle, and the forearm on the extensor digitorum. The examiner applied gradual pressure on the defined areas, and patients were asked to report the exact moment when the pressure began to change to a sensation of pain. At that time, the examiner terminated the application of pressure, and the measurement related to the PPT was taken.

Kinematic parameters were analyzed by two functional tests, the 10-Meter Walking Test (10MWT) and the Time Up&Go test (TUG). The tests were carried out with the help of an inertial sensor (BTS G-Sensor), placed at the trunk level, above the subject's clothing, via an elastic belt. 10MWT is a standard test used in gait assessment that consists of walking 10 meters in a straight line; TUG is a common and validated test that provides important indications about the level of balance and functional and walking ability of subjects. The test consists of getting up from a chair, walking 3 meters, turning around, returning to the chair, and sitting down. The inertial sensor registered the spatio-temporal parameters during 10MWT and TUG.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for this study are age 50 and 90 years, Body Mass Index (BMI) <30 kg/m2, and Knee OA symptoms. OA is confirmed by the treating physician and radiographic findings (severity of OA 2 to 4 Kellgren-Lawrence scale).

Exclusion Criteria:

Exclusion Criteria are the presence of psychiatric or neurological disorders, peripheral nerve injury, uncontrolled inflammatory states, neuromuscular and rheumatologic diseases, dementia and language barriers, limiting orthopedic conditions (amputations, non-reducible joint limitations), post-traumatic OA (e.g., fractures), congenital hip deformities, hip surgery, Legg-Calvé-Perthes disease. Patients with degenerative or non-degenerative neurological conditions in which pain perception is impaired and ongoing corticosteroid infiltration, and bedridden subjects are excluded.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to clinic IRCCS Fondazione Don Carlo Gnocchi, Italy diagnosed with knee OA will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
WOMAC scale | Single assessment at baseline
  a patient-reported outcome questionnaire that aims to identify changes in symptoms and activity restrictions in subjects with OA.

SECONDARY OUTCOMES:
Pain DETECT Scale | Single assessment at baseline
  The PainDETECT questionnaire (PD-Q) is a screening instrument designed to classify whether a patient has neuropathic pain.
Central Sensitization Inventory (CSI) Index | Single assessment at baseline
  The Central Sensitisation Inventory (CSI) is a self-report outcome measure designed to identify patients with symptoms related to central sensitization.
Patient Health Questionairre (PHQ-9) | Single assessment at baseline
post traumatic distress checklist (PTSD) | Single assessment at baseline
  The PCL-5 is a 20-item self-report checklist of PTSD symptoms based closely on the DSM-5 criteria.
Pain Catastrophyzing Scale (PCS) | Single assessment at baseline
  The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking due to pain according to 3 components: rumination, magnification, and helplessness.
Tampa Kinesiophobia Scale (TSK) | Single assessment at baseline
  The Tampa Scale for Kinesiophobia (TSK) is a 17-item questionnaire that quantifies fear of movement.
Fear Avoidance Believe Questionnaire (FABQ) | Single assessment at baseline
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient-reported questionnaire that specifically focuses on a patient's fear avoidance beliefs.
Injustice Experience Questionnaire (IEQ) | Single assessment at baseline
  he Injustice Experience Questionnaire (IEQ) assesses the degree to which chronic pain sufferers perceive injustice in relation to their pain.
10 meters walking test | Single assessment at baseline
  10MWT is a standard test used in gait assessment that consists of walking 10 meters in a straight line.
Time up and Go test | Single assessment at baseline
  TUG is a common and validated test that provides important indications about the level of balance and functional and walking ability of subjects. The test consists of getting up from a chair, walking 3 meters, turning around, returning to the chair, and sitting down.
Pressure pain threshold assessment | Single assessment at baseline
  An assessment of pressure pain threshold (PPT) was conducted through an electronic algometer (Algomed)17. The defined sites for PPT were the patella, Gerdy's tubercle, and the forearm on the extensor digitorum. The examiner applied gradual pressure on the defined areas, and patients were asked to report the exact moment when the pressure began to change to a sensation of pain. At that time, the examiner terminated the application of pressure, and the measurement related to the PPT was taken.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Italy, Rovato, Italy

IPD SHARING:
Plan to Share IPD: No